CLINICAL TRIAL: NCT03023423
Title: A Phase 1b/2, Open-Label, Randomized Study of Daratumumab Administered in Combination With Atezolizumab Compared With Atezolizumab Alone in Subjects With Previously Treated Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Daratumumab in Combination With Atezolizumab Compared With Atezolizumab Alone in Participants With Previously Treated Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: DARZALEX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108256; 2016-002579-83 (EudraCT Number); 54767414LUC2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-12-09; First posted 2017-01-18 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A: Atezolizumab (Experimental): Participants in Treatment Arm A will receive Atezolizumab 1,200 milligram (mg) intravenously (IV) on Day 1 of every 21-day cycle. Participants with confirmed disease progression based on RECIST 1.1 may cross over to Arm B and receive daratumumab and atezolizumab, provided crossover eligibility criteria are met.
  Interventions: Drug: Atezolizumab
- Treatment Arm B: Atezolizumab and Daratumumab (Experimental): Participants will receive daratumumab 16 milligram per kilogram [mg/kg] (Safety Run-in and Treatment Arm B) Intravenously (IV) weekly for 3 cycles (Day 1, 8 and 15), and Day 1 of every 21-day cycle thereafter. Atezolizumab will be administered at 1200 mg IV on Day 2 of Cycle 1 and on Day 1 of every 21-day cycle thereafter. Participants will continue to receive study treatment until confirmed disease progression, unacceptable toxicity, or any other treatment discontinuation criteria are met.
  Interventions: Drug: Atezolizumab; Drug: Daratumumab

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive atezolizumab 1200 mg intravenously.
Drug: Daratumumab — Participants will receive daratumumab 16 mg/kg intravenously.
  Other Names: JNJ-54767414
  Arms: Treatment Arm B: Atezolizumab and Daratumumab

SUMMARY:
The purpose of the study is to compare the overall response rate (ORR) in non-small cell lung cancer (NSCLC) participants treated with daratumumab in combination with atezolizumab versus atezolizumab alone.

DETAILED DESCRIPTION:
This randomized (study medication assigned to participants by chance), multicenter study will provide study treatment (atezolizumab alone or atezolizumab+daratumumab) to participants with previously treated advanced or metastatic NSCLC to assess the anti-tumor activity and safety. Participants who receive atezolizumab treatment with confirmed disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 will be eligible to crossover to treatment (atezolizumab + daratumumab) if they meet crossover eligibility criteria. It is expected that 100 participants will enroll in the study including 6 participants in the safety run in phase. Data Monitoring Committee (DMC) will review ongoing data, and may formulate recommendations on study conduct, including expansion of enrollment of some PD-L1 subgroups, resulting in greater than 96 participants. The participants in the safety run in phase will be administered the combination of daratumumab and atezolizumab to determine the safety and tolerability that will be evaluated by the Safety Evaluation Team (SET) for dose limiting toxicity before the random assignment of participants in a 1:1 ratio in 2 treatment arms. The study consists of 3 phases: Screening Phase (up to 28 days), Treatment Phase and Post-Treatment Follow-up Phase which will continue until death, lost to follow-up, withdrawal of consent, or the End of the Study [the study end is approximately 6 to 12 months after that last participant is enrolled]. Participants will undergo tumor assessments (RECIST 1.1), immunogenicity, pharmacokinetics, biomarkers and safety evaluations (adverse events, laboratory tests, electrocardiogram [ECGs], vital sign measurements, physical examinations, Eastern Cooperative Oncology Group [ECOG] performance status score) over the time.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have histologically or cytologically confirmed advanced or metastatic non-small cell lung cancer (NSCLC) (Stage IIIb or greater)
* Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Tumor cell programmed death-ligand 1 (PD-L1) score of tumor cells (TC)1-3 and immune cell PD-L1 score of tumor-infiltrating immune cells (IC)0-3 as determined by an immunohistochemistry (IHC) assay performed by the central laboratory on tissue obtained after the last line of therapy
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta- hCG]) at Screening within 14 days prior to study drug administration

Inclusion Criteria for Crossover:

* Participants must have been randomized to Arm A of the study and had radiographic disease progression according to RECIST 1.1
* Participants must have a mandatory biopsy at the time of disease progression according to RECIST 1.1 prior to crossing over. If not clinically feasible, discussion with Sponsor is required
* The first dose of atezolizumab in the crossover arm should be within 42 days of last dose but no less than 21 days from the last dose prior to crossing over

Exclusion Criteria:

* Received any of the following prescribed medications or therapies in the past:

  1. Anti-cluster of differentiation(CD)38 therapy, including daratumumab
  2. CD137 agonists, immune checkpoint inhibitors including but not limited to CTLA-4, anti-PD-1, and anti-PD-L1 therapies
* Known to be seropositive for human immunodeficiency virus (HIV)
* Prior allogeneic bone marrow transplantation or solid organ transplant
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Active hepatitis B, defined by a positive test for hepatitis B surface antigen [HBsAg] or prior history of hepatitis B, defined by presence of antibodies to hepatitis B core antigen [anti-HBc], regardless of hepatitis B surface antibody [anti-HBs] status; active hepatitis C or prior history of hepatitis C (anti-HCV positive), except in the setting of a sustained virologic response (SVR), defined as aviremia 12 weeks after completion of antiviral therapy. If hepatitis C virus (HCV) antibodies are detected, an HCV RNA test for viral load by polymerase chain reaction (PCR) should be performed at least 12 weeks after completion of antiviral therapy to rule out active infection

Exclusion Criteria for Crossover:

* Received any subsequent anti-cancer therapies from the time between the last dose of atezolizumab prior to the first administration of study drug after crossing over
* Whole brain radiation within 28 days or other radiotherapy within 14 days prior to first administration of study drug after crossing over

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (47):
- United States (16):
  - Loma Linda, California
  - Whittier, California
  - Newark, Delaware
  - Deerfield Beach, Florida
  - Fort Lauderdale, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - New Orleans, Louisiana
  - Bethesda, Maryland
  - Oklahoma City, Oklahoma
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Spokane, Washington
- France (12):
  - Bordeaux
  - Boulogne-Billancourt
  - Caen
  - Créteil
  - Haut-Rhin
  - Montpellier
  - Nancy
  - Paris
  - Rennes
  - Rouen
  - Suresnes
  - Vandœuvre-lès-Nancy
- Hungary (3):
  - Budapest
  - Székesfehérvár
  - Tatabánya
- Poland (3):
  - Lodz
  - Otwock
  - Wieliszew
- Spain (13):
  - Barcelona
  - Elche
  - Jaén
  - Leganés
  - Madrid
  - Málaga
  - Murcia
  - Palma de Mallorca
  - Pozuelo de Alarcón
  - San Sebastián
  - Sótano
  - Valencia
  - Zaragoza

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 100 participants were enrolled in the study (7 in phase 1b [safety run-in phase], and 93 in Phase 2 [randomized phase]). Among them, 99 participants (7 in phase 1b [safety run-in phase], and 92 in phase 2 [randomized phase]) were randomized as 1 participant was randomized after the clinical cutoff date (17-May-2018).
Groups:
- Safety Run-in Phase: Daratumumab + Atezolizumab: Participants received daratumumab (Dara) 16 milligram per kilogram (mg/kg) intravenously (IV) weekly on Days 1, 8, and 15 for first 3 cycles and then on Day 1 of each 21-day cycle thereafter along with atezolizumab (Atezo) IV at a dose of 1200 milligram (mg) on Day 2 of Cycle 1 and on Day 1 of every 21-day cycle thereafter until disease progression, unacceptable toxicity or other protocol-defined treatment discontinuation criteria.
- Randomized Phase: Atezolizumab: Participants received atezolizumab IV at a dose of 1200 milligram (mg) on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity or other protocol-defined treatment discontinuation criteria.
- Randomized Phase: Daratumumab + Atezolizumab: Participants received daratumumab 16 mg/kg IV weekly on Days 1, 8, and 15 for first 3 cycles and then on Day 1 of each 21-day cycle thereafter along with atezolizumab IV at a dose of 1200 mg on Day 2 of Cycle 1 and on Day 1 of every 21-day cycle thereafter until disease progression, unacceptable toxicity or other protocol-defined treatment discontinuation criteria.
Period: Overall Study
Arm/Group | Safety Run-in Phase: Daratumumab + Atezolizumab | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab
Started | 7 | 46 | 46
Treated | 7 | 44 | 44
Crossover From Atezo to Dara + Atezo | 0 | 8 (Participants who met crossover eligibility criteria entered to Dara + Atezo arm.) | 0
Completed | 0 | 0 | 0
Not Completed | 7 | 46 | 46
Not completed — Death | 5 | 12 | 20
Not completed — Other | 0 | 2 | 2
Not completed — Ongoing | 2 | 32 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run-in Phase: Daratumumab + Atezolizumab | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab | Total
Number analyzed (Participants) | 7 | 46 | 46 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9.73) | 61.7 (10.05) | 63.2 (10.76) | 62.3 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 18 | 8 | 29
  Male | 4 | 28 | 38 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 36 | 40 | 83
  Unknown or Not Reported | 0 | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 35 | 41 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 11 | 5 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Other | 0 | 11 | 6 | 17
  White Non-Hispanic | 7 | 35 | 40 | 82
Region of Enrollment [Count of Participants; unit: Participants]
  FRANCE | 0 | 10 | 6 | 16
  HUNGARY | 0 | 8 | 7 | 15
  SPAIN | 3 | 19 | 27 | 49
  UNITED STATES | 4 | 9 | 6 | 19
Time from initial diagnosis [Mean (Standard Deviation); unit: months] — Time from initial diagnosis is defined as the time from the initial diagnosis of non-small cell lung cancer (NSCLC) to the first dosing date or randomization date (if first dosing date is missing).
  months | 10.3 (9.29) | 18.8 (20.89) | 17.6 (14.17) | 17.6 (17.37)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status was used to evaluate the effect of the disease status on the activities of daily living. ECOG performance status was determined by ECOG 5-point scale: 0=Fully active, 1=Ambulatory, carry out work of sedentary nature, 2=Ambulatory, capable of all self-care, 3=Capable of limited self-care, confined to bed or chair more than 50% of waking hours, 4=Completely disabled, no self-care, totally confined to bed or chair, 5=Dead.
  Participants
    ECOG Score 0 | 3 | 19 | 12 | 34
    ECOG Score 1 | 4 | 27 | 33 | 64
    ECOG Score 2 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with partial response (PR) or complete response (CR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Criteria for CR: Disappearance of all target lesions; all lymph nodes must be of non-pathological in size (less than [<]10 millimeter [mm] short axis; normalization of tumor marker level. Criteria for PR: greater than or equal to (>=)30 percent (%) decrease in sum of the diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. Overall Response (OR) = CR + PR. The outcome measure (OM) was planned to be reported for participants based on their initial assignment to Randomized Phase: Atezolizumab'.
Time Frame: Up to 1.5 years
Population: Intent-to-treat (ITT) analysis set included all participants who had entered the Randomized phase of the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 46 | 46
Percentage of participants | 13.0 [4.9 to 26.3] | 4.3 [0.5 to 14.8]
Statistical Analysis 1: Comparison: Randomized Phase: Atezolizumab vs Randomized Phase: Daratumumab + Atezolizumab; Test type: Superiority; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.03 to 1.92]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Crossover participants were counted twice (in 'Randomized Phase: Atezo arm' and in 'Randomized Phase: Atezo Crossed Over to Dara + Atezo') for safety analysis. For cross-over participants, AEs after initiation of cross-over treatment were summarized separately in the crossover arm, however, AEs occurred before crossover treatment were included in 'Randomized Phase: Atezolizumab arm'.
Time Frame: Up to 1.5 years
Population: Safety analysis set included all participants who had received at least 1 administration of any study medication.
Measure: Number; unit: Participants
Groups:
- Safety Run-in: Atezolizumab + Daratumumab: Participants received daratumumab 16 milligram per kilogram (mg/kg) Intravenously (IV) weekly for first 3 cycles and every 3 weeks for all cycles thereafter along with atezolizumab IV at a dose of 1200 milligram (mg) on Day 2 of Cycle 1 and on Day 1 of every 21-day cycle thereafter.
- Randomized Phase: Atezo Crossed Over to Dara + Atezo: Participants who crossed over from Atezolizumab arm (Randomized Phase) to Daratumumab + Atezolizumab arm (Randomized Phase) received daratumumab 16 mg/kg IV weekly on Days 1, 8, and 15 for first 3 cycles and then on Day 1 of each 21-day cycle thereafter along with atezolizumab IV at a dose of 1200 mg on Day 2 of Cycle 1 and on Day 1 of every 21-day cycle thereafter until disease progression, unacceptable toxicity or other protocol defined treatment discontinuation criteria.
Arm/Group | Safety Run-in: Atezolizumab + Daratumumab | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab | Randomized Phase: Atezo Crossed Over to Dara + Atezo
Number analyzed (Participants) | 7 | 44 | 44 | 8
Participants | 7 | 42 | 44 | 8

3. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response was defined as duration from date of initial documentation of disease response to date of first objectively documented evidence of recurrence or progressive disease (PD) or death, whichever occurred first. PD: Sum of diameters increased by >=20% and >=5 millimeter (mm) from nadir (including baseline if it was smallest sum). Participants with measurable disease: for "unequivocal progression" based on non-target disease, overall level of substantial worsening that merits discontinuation of therapy (if target disease was stable disease [SD]/PR). Participants without measurable disease: for "unequivocal progression" of non-target disease, increase in overall tumor burden comparable to increase required for PD of measurable disease. Appearance of 1/ more new lesions or unequivocal progression of non-target lesion was also considered as PD. The OM was planned to be reported for participants based on their initial assignment to 'Randomized Phase: Atezolizumab'.
Time Frame: Up to 1.5 years
Population: ITT analysis set included all participants who had entered the Randomized phase of the study. Here, N (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 6 | 2
Months | 5.8 [2.2 to 5.8] | 2.9 [NA to NA] — Here NA signifies that the lower and upper limit of 95% Confidence Interval (CI) were not estimable due to lesser number of participants with events.

4. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate was defined as percentage of participants who achieved disease control (CR, PR, or SD). RECIST 1.1 Criteria for CR: Disappearance of all target lesions; all lymph nodes of non-pathological in size (<10 mm short axis); normalization of tumor marker level. Criteria for PR: >=30 % decrease in sum of the diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. Criteria for SD: <30% decrease in sum of diameters of all target lesions compared with baseline and <20% increase compared with nadir, in absence of new lesions or unequivocal progression of nontarget lesions. The OM was planned to be reported for participants based on their initial assignment to 'Randomized Phase: Atezolizumab'.
Time Frame: Up to 1.5 years
Population: ITT analysis set included all participants who had entered the Randomized phase of the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 46 | 46
Percentage of Participants | 43.5 [28.9 to 58.9] | 52.2 [36.9 to 67.1]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the duration from the date of randomization until the first documented disease progression (PD) or death, whichever occurred first. PD: Sum of diameters increased by >=20% and >=5 millimeter (mm) from nadir (including baseline if it was smallest sum). Participants with measurable disease: for "unequivocal progression" based on non-target disease, overall level of substantial worsening that merits discontinuation of therapy (if target disease was stable disease [SD]/PR). Participants without measurable disease: for "unequivocal progression" of non-target disease, increase in overall tumor burden comparable to increase required for PD of measurable disease. Appearance of 1/ more new lesions or unequivocal progression of non-target lesion was also considered as PD. The OM was planned to be reported for participants based on their initial assignment to 'Randomized Phase: Atezolizumab'.
Time Frame: Up to 1.5 years
Population: ITT analysis set included all participants who had entered the Randomized phase of the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 46 | 46
Months | 1.48 [1.38 to 2.76] | 1.68 [1.41 to 2.79]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the duration from the date of randomization to the date of participant's death due to any cause. The OM was planned to be reported for participants based on their initial assignment to 'Randomized Phase: Atezolizumab'.
Time Frame: Up to 1.5 years
Population: ITT analysis set included all participants who had entered the Randomized phase of the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 46 | 46
Months | NA [7.43 to NA] — Here NA signifies that the median and upper limit of 95% CI were not estimable due to lesser number of events. | 7.13 [3.52 to NA] — Here NA signifies that the upper limit of 95% CI was not estimable due to lesser number of events.

7. Secondary Outcome: Daratumumab Serum Concentration
Description: Daratumumab serum concentrations were reported. Each cycle was of 21-days. The OM was planned to be reported for participants based on their initial assignment to 'Randomized Phase: Atezolizumab'.
Time Frame: Cycle 1 Day 1 (C1D1):predose and postdose; C2D1 and C3D1:predose; C3D15: predose and postdose; C4D1: predose and postdose; C8D1: predose and postdose; C12D1: predose; end of treatment (37 days after last dose); and post last dose (up to 1.5 years)
Population: Pharmacokinetic (PK)-evaluable analysis set included all participants who had received at least 1 dose of daratumumab or atezolizumab and had at least 1 postinfusion sample collected. Here 'n' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure at a given time point.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Safety Run-in: Atezolizumab + Daratumumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 7 | 43
Microgram per milliliter (mcg/mL)
  Cycle 1 Day 1 Predose | 0.00 (0.000) | 0.00 (0.000)
  Cycle 1 Day 1 Postdose: number analyzed (Participants) | 6 | 38
  Cycle 1 Day 1 Postdose | 417.13 (141.626) | 296.12 (85.660)
  Cycle 2 Day 1 Predose: number analyzed (Participants) | 4 | 35
  Cycle 2 Day 1 Predose | 393.95 (139.480) | 278.42 (89.340)
  Cycle 3 Day 1 Predose: number analyzed (Participants) | 3 | 26
  Cycle 3 Day 1 Predose | 740.17 (99.515) | 487.65 (124.935)
  Cycle 3 Day 15 Predose: number analyzed (Participants) | 4 | 24
  Cycle 3 Day 15 Predose | 843.22 (156.792) | 552.79 (180.549)
  Cycle 3 Day 15 Postdose: number analyzed (Participants) | 4 | 23
  Cycle 3 Day 15 Postdose | 1088.73 (282.349) | 827.72 (266.085)
  Cycle 4 Day 1 Predose: number analyzed (Participants) | 3 | 22
  Cycle 4 Day 1 Predose | 899.90 (123.305) | 574.81 (181.193)
  Cycle 4 Day 1 Postdose: number analyzed (Participants) | 3 | 21
  Cycle 4 Day 1 Postdose | 1416.40 (353.415) | 856.30 (244.698)
  Cycle 8 Day 1 Predose: number analyzed (Participants) | 1 | 8
  Cycle 8 Day 1 Predose | 254.87 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant. | 288.84 (177.187)
  Cycle 8 Day 1 Postdose: number analyzed (Participants) | 1 | 8
  Cycle 8 Day 1 Postdose | 824.64 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant. | 617.21 (239.962)
  Cycle 12 Day 1 Predose: number analyzed (Participants) | 0 | 2
  Cycle 12 Day 1 Predose |  | 260.21 (17.163)
  End of Treatment: number analyzed (Participants) | 3 | 13
  End of Treatment | 405.14 (242.189) | 187.75 (110.531)
  Post Last Dose: number analyzed (Participants) | 2 | 5
  Post Last Dose | 41.84 (23.082) | 112.63 (115.727)

8. Secondary Outcome: Atezolizumab Serum Concentration
Description: Atezolizumab serum concentrations were reported. Each cycle was of 21-days. The OM was planned to be reported for participants based on their initial assignment to 'Randomized Phase: Atezolizumab'.
Time Frame: C1D1:predose and postdose; C1D2:predose and postdose; C2D1, C3D1:predose; C3D15:predose and postdose; C4D1:predose and postdose; C8D1:predose and postdose; C12D1:predose; end of treatment (37 days after last dose); and post last dose (up to 1.5 years)
Population: PK-evaluable analysis set: all participants who received at least 1 dose of daratumumab/atezolizumab and had at least 1 postinfusion sample collected. Here N (number of participants analyzed): participants evaluable for this outcome measure, and n (number of participants analyzed): participants evaluable for this outcome measure at given timepoint.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Safety Run-in: Atezolizumab + Daratumumab | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 7 | 39 | 39
Microgram per milliliter (mcg/mL)
  Cycle 1 Day 1 Predose: number analyzed (Participants) | 0 | 37 | 13
  Cycle 1 Day 1 Predose |  | 0.00 (0.000) | 0.00 (0.000)
  Cycle 1 Day 1 Postdose: number analyzed (Participants) | 0 | 37 | 3
  Cycle 1 Day 1 Postdose |  | 396.51 (103.196) | 440.00 (93.145)
  Cycle 1 Day 2 Predose: number analyzed (Participants) | 7 | 0 | 24
  Cycle 1 Day 2 Predose | 0.00 (0.000) |  | 0.00 (0.000)
  Cycle 1 Day 2 Postdose: number analyzed (Participants) | 7 | 0 | 34
  Cycle 1 Day 2 Postdose | 362.14 (43.434) |  | 343.82 (135.476)
  Cycle 2 Day 1 Predose: number analyzed (Participants) | 5 | 30 | 20
  Cycle 2 Day 1 Predose | 91.16 (15.305) | 78.85 (30.575) | 81.90 (20.021)
  Cycle 3 Day 1 Predose: number analyzed (Participants) | 2 | 21 | 17
  Cycle 3 Day 1 Predose | 176.50 (33.234) | 117.61 (33.227) | 123.51 (31.882)
  Cycle 4 Day 1 Predose: number analyzed (Participants) | 2 | 18 | 12
  Cycle 4 Day 1 Predose | 166.50 (37.477) | 145.64 (37.323) | 157.79 (37.819)
  Cycle 4 Day 1 Postdose: number analyzed (Participants) | 4 | 17 | 18
  Cycle 4 Day 1 Postdose | 612.25 (81.578) | 539.24 (116.291) | 482.33 (139.879)
  Cycle 8 Day 1 Predose: number analyzed (Participants) | 0 | 6 | 0
  Cycle 8 Day 1 Predose |  | 158.23 (77.778) |
  Cycle 8 Day 1 Postdose: number analyzed (Participants) | 0 | 8 | 4
  Cycle 8 Day 1 Postdose |  | 527.50 (213.492) | 515.25 (214.177)
  Cycle 12 Day 1 Predose: number analyzed (Participants) | 0 | 1 | 1
  Cycle 12 Day 1 Predose |  | 183.00 (NA) — Here NA signifies that the standard deviation could not be calculated for a single participant. | 248.00 (NA) — Here NA signifies that the standard deviation could not be calculated for a single participant.
  End of Treatment: number analyzed (Participants) | 3 | 11 | 12
  End of Treatment | 136.43 (73.002) | 129.55 (79.720) | 141.62 (71.756)
  Post Last Dose: number analyzed (Participants) | 1 | 2 | 2
  Post Last Dose | 33.10 (NA) — Here NA signifies that the standard deviation could not be calculated for a single participant. | 13.17 (8.386) | 115.10 (146.937)

9. Secondary Outcome: Number of Participants With Anti-Daratumumab Antibodies
Description: Number of participants with antibodies to daratumumab (tested using a validated immunoassay method) were reported. The OM was planned to be reported for participants based on their initial assignment to 'Randomized Phase: Atezolizumab'.
Time Frame: Up to 1.5 years
Population: The immunogenicity-evaluable analysis set included all participants who received at least 1 dose of atezolizumab or daratumumab and had appropriate samples for detection of antibodies to atezolizumab or daratumumab. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Safety Run-in: Atezolizumab + Daratumumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 7 | 37
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Anti-Atezolizumab Antibodies
Description: Number of participants with antibodies to atezolizumab (tested using a validated immunoassay method) were reported. The OM was planned to be reported for participants based on their initial assignment to 'Randomized Phase: Atezolizumab'.
Time Frame: Up to 1.5 years
Population: The immunogenicity-evaluable analysis set included all participants who received at least 1 dose of atezolizumab or daratumumab and had appropriate samples for detection of antibodies to atezolizumab or daratumumab.
Measure: Number; unit: Participants
Arm/Group | Safety Run-in: Atezolizumab + Daratumumab | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab
Number analyzed (Participants) | 7 | 39 | 38
Participants | 0 | 6 | 5

ADVERSE EVENTS:
Time Frame: Up to 1.5 years
Description: Safety analysis set included participants who received at least 1 administration of any study medication. Crossover participants were counted twice (in 'Randomized Phase: Atezo arm' and 'Randomized Phase: Atezo Crossed Over to Dara + Atezo') for safety analysis. For cross-over participants, adverse events (AEs) after initiation of cross-over treatment summarized separately in crossover arm, however, AEs occurred before crossover treatment were included in 'Randomized Phase: Atezolizumab arm'.
Groups:
- Randomized Phase: Atezo Crossed Over to Dara + Atezo: Participants who crossed over from Atezolizumab arm (Randomized Phase) to Daratumumab + Atezolizumab arm (Randomized Phase) received daratumumab 16 mg/kg IV weekly on Days 1, 8, and 15 for first 3 cycles and then on Day 1 of each 21-day cycle thereafter along with atezolizumab IV at a dose of 1200 mg on Day 2 of Cycle 1 and on Day 1 of every 21-day cycle thereafter until disease progression, unacceptable toxicity or other protocol-defined treatment discontinuation criteria.
Arm/Group | Safety Run-in Phase: Daratumumab + Atezolizumab | Randomized Phase: Atezolizumab | Randomized Phase: Daratumumab + Atezolizumab | Randomized Phase: Atezo Crossed Over to Dara + Atezo
All-Cause Mortality (participants affected / at risk) | 5/7 | 9/44 | 20/44 | 3/8
Serious Adverse Events (participants affected / at risk) | 4/7 | 15/44 | 21/44 | 3/8
Other Adverse Events (participants affected / at risk) | 7/7 | 41/44 | 41/44 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Phase: Daratumumab + Atezolizumab (N=7) | Randomized Phase: Atezolizumab (N=44) | Randomized Phase: Daratumumab + Atezolizumab (N=44) | Randomized Phase: Atezo Crossed Over to Dara + Atezo (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1 | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 1 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0
Sudden Death (General disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Oral Infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 3 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 3 | 0
Superinfection (Infections and infestations) | 0 | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bronchial Fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Phase: Daratumumab + Atezolizumab (N=7) | Randomized Phase: Atezolizumab (N=44) | Randomized Phase: Daratumumab + Atezolizumab (N=44) | Randomized Phase: Atezo Crossed Over to Dara + Atezo (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 6 | 7 | 1
Sinus Tachycardia (Cardiac disorders) | 2 | 0 | 2 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 3 | 0 | 0
Dry Eye (Eye disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 6 | 0
Constipation (Gastrointestinal disorders) | 2 | 5 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 4 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 8 | 7 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 6 | 1
Asthenia (General disorders) | 3 | 15 | 14 | 2
Chest Discomfort (General disorders) | 2 | 0 | 2 | 0
Chest Pain (General disorders) | 0 | 3 | 3 | 2
Chills (General disorders) | 1 | 0 | 3 | 1
Fatigue (General disorders) | 3 | 7 | 9 | 2
Malaise (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 5 | 4 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 4 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 7 | 11 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 8 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 1
Headache (Nervous system disorders) | 3 | 2 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 3 | 2 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 16 | 3
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 13 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 5 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 1
Flushing (Vascular disorders) | 1 | 0 | 2 | 0
Hypertension (Vascular disorders) | 4 | 0 | 4 | 0
Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 1
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0
Localised Oedema (General disorders) | 0 | 0 | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 1 | 1
Oedema Peripheral (General disorders) | 0 | 2 | 2 | 0
Pain (General disorders) | 0 | 2 | 0 | 1
Secretion Discharge (General disorders) | 0 | 0 | 1 | 0
Temperature Intolerance (General disorders) | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 2 | 0
Buttock Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 2 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 2 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1 | 0 | 0
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 0 | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 0 | 1 | 1 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 1 | 0
Weight Increased (Investigations) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 2 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Vein Thrombosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hair Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT03023423/SAP_000.pdf
  • Study Protocol (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT03023423/Prot_001.pdf